CLINICAL TRIAL: NCT04250116
Title: Appropriate Duration of Anti-Platelet and Thrombotic Strategy After 12 Months in Patients With Atrial Fibrillation Treated With Drug Eluting Stents (ADAPT AF-DES)
Brief Title: Appropriate Duration of Anti-Platelet and Thrombotic Strategy After 12 Months in Patients With Atrial Fibrillation Treated With Drug Eluting Stents
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-1128
Record Dates: First submitted 2020-01-19; First posted 2020-01-31 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — N(4)-oleylcytosine arabinoside; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOAC monotherapy (Experimental)
  Interventions: Drug: NOAC monotherapy
- Dual antithrombotic therapy (Active Comparator)
  Interventions: Drug: Dual antithrombotic therapy with NOAC and clopidogrel

INTERVENTIONS:
Drug: NOAC monotherapy — Patients enrolled in the NOAC monotherapy arm would be administered with apixaban 5 mg twice daily or rivaroxaban 20 mg once daily for 2 years after randomization. Reduced dose of apixaban (2.5 mg twice daily) or rivaroxaban (15 mg once daily) will be used in patients meeting the pre-defined criteria for dose reduction. Warfarin is allowed to use at the physicians' discretion.
  Arms: NOAC monotherapy
Drug: Dual antithrombotic therapy with NOAC and clopidogrel — Patients enrolled in the dual antithrombotic therapy arm would be administered with apixaban 5 mg twice daily or rivaroxaban 15 mg once daily and clopidogrel 75 mg daily for 2 years after randomization. Reduced dose of apixaban (2.5 mg twice daily) or rivaroxaban (10 mg once daily) will be used in patients meeting the pre-defined criteria for dose reduction. Warfarin is allowed to use at the physicians' discretion.
  Arms: Dual antithrombotic therapy

SUMMARY:
Atrial fibrillation patients with risk factors for stroke and systemic embolism require long-term anticoagulant therapy. Recently, non-vitamin K antagonist oral anticoagulant (NOAC) has shown their excellent safety and efficacy, and thus are widely accepted in clinical practice. Meanwhile, after percutaneous coronary intervention (PCI) using the drug-eluting stents due to coronary artery disease, the administration of one or more antiplatelets is essential to prevent the recurrence of stent thrombosis and myocardial infarction. Combined administration of anticoagulants and antiplatelets significantly lowers the incidence of ischemic events such as stroke and myocardial infarction, however, it also significantly increases the likelihood of bleeding leading to hospitalization, and or even death, thereby significantly affecting the clinical course of the AF patients who underwent PCI. Nevertheless, due to the very high mortality rate of stent thrombosis, the current standard of care guidelines recommend triple therapy with anticoagulants and double antiplatelet therapy (DAPT) in patients with atrial fibrillation for 1 month after coronary intervention, followed by co-administration of NOAC with single antiplatelet agent for 1 year. However, little is known after the optimal therapeutic strategy after 1 year. The purpose of this study is to compare the clinical results of single anticoagulant and clopidogrel combination therapy for maintenance therapy after 1 year in patients with atrial fibrillation.

DETAILED DESCRIPTION:
AF patients who had undergone PCI with DES implantation at least 12 months ago will be enrolled in this study. Decision for the antiplatelet agent discontinuation would be determined by randomization. Apixaban or Rivaroxaban would be prescribed to reduce the risk stroke or systemic embolism evoked by AF, and the administration of Warfarin, a vitamin-K dependent anticoagulant, would also be allowed according to attending physician's decision. The following criteria should be followed for the reduction of dosages according to the patient's renal function and other systemic conditions. Warfarin is administered to patients with creatinine clearance < 15 ml/min or dialysis. The drugs used in this study correspond to the international treatment guidelines after coronary intervention in patients with atrial fibrillation.NOAC and antiplatelet agents would be prescribed upon an outpatient visit. Clinical outcome would be followed for 2 years after study enrollment and randomization.

Screening

* Baseline Serum AST/ALT level
* Creatinine clearance (mL/min)
* Concurrent administration of CYP3A4 agents: Ketoconazole, Itraconazole, Iopinavir/ritonavir, indinavir/ritonavir, conviaptan

  # Dose Adjustment Criteria for Apixaban

  @ Meeting 2 of 3 following criteria
* Serum creatinine level > 1.5 mg/dL
* Body weight under 60 kg
* age over 80 years old

  # Dose Adjustment Criteria for Rivaroxaban
* eGFR from 15-49 mg/min

ELIGIBILITY:
Inclusion Criteria:

1. over 19 years old
2. Patient who underwent PCI with DES more than 12 months ago
3. Non-valvular atrial fibrillation patients requiring long-term anticoagulation

Exclusion Criteria:

1. Over 85 years old
2. Pregnancy or Potential Pregnancy
3. Life expectancy within 1 year
4. Patients who refuse or do not understand the written consent form
5. Requiring anticoagulation due to history of mechanical valve replacement, mitral stenosis or deep vein thrombosis
6. Coagulopathy, continuous bleeding, or Hb level below 10 g/dL
7. Intracerebral hemorrhage within 2 months
8. Patients with gastrointestinal hemorrhage within three months of registration
9. Patients diagnosed with a gastrointestinal tumor that requires continuous treatment
10. Patients treated with 1st generation drug-eluting stents (Cypher, Taxus, or Endeavor Sprint)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical event (NACE) | at 12 months (1 year)
  All-cause death, myocardial infarction, stent thrombosis, stroke, systemic embolism, major or clinically relevant non-major bleeding defined by International Society on Thrombosis and Haemostasis (ISTH)

SECONDARY OUTCOMES:
Each component of NACE | Day 1 to 12 months (1 year)
  1) all-cause death; 2) myocardial infarction; 3) stent thrombosis; 4) stroke; 5) systemic embolism; 6) ISTH major bleeding; 7) ISTH clinically relevant non-major bleeding
ISTH major or clinically relevant non-major bleeding | Day 1 to 12 months (1 year)
All-cause death, myocardial infarction, stent thrombosis, stroke, systemic embolism, and ISTH major bleeding | Day 1 to 12 months (1 year)
Cardiovascular death | Day 1 to 12 months (1 year)
Cardiovascular death, myocardial infarction, stent thrombosis, ischemic stroke, and systemic embolism | Day 1 to 12 months (1 year)
Primary outcome (NACE) at 2 years | Day 1 to 24 months (2 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SJ, Yu HT, Lee YJ, Lee SH, Heo JH, Ahn SG, Shin S, Doh JH, Her AY, Cho BR, Kim GS, Kwon TG, Lim SW, Shim J, Jang JY, Lee K, Cho YH, Choi CU, Lee SR, Park HB, Lee HC, Kim S, Yun KH, Ahn JH, Lee BK, Cho DK, Kim SY, Kim U, Kang TS, Choi SH, Kim WH, Lee JB, Rhee MY, Kim JB, Jo SH, Hyun DW, Kim D, Kim TH, Hong SJ, Uhm JS, Shin DH, Ahn CM, Kim BK, Joung B, Ko YG, Choi D, Hong MK, Jang Y, Pak HN, Kim JS; ADAPT AF-DES Investigators. Therapy for Atrial Fibrillation in Patients with Drug-Eluting Stents. N Engl J Med. 2025 Nov 8. doi: 10.1056/NEJMoa2512091. Online ahead of print. PMID 41211917
- [Derived] Lee SH, Lee SJ, Heo JH, Ahn SG, Doh JH, Shin S, Shim J, Her AY, Kim BG, Lim SW, Kwon TG, Lee KH, Kim D, Lee YJ, Yu HT, Kim TH, Shin DH, Pak HN, Kim JS. Optimal antithrombotic strategy in patients with atrial fibrillation beyond 1 year after drug-eluting stent implantation: Design and rationale of the randomized ADAPT AF-DES trial. Am Heart J. 2024 May;271:48-54. doi: 10.1016/j.ahj.2024.02.014. Epub 2024 Feb 23. PMID 38401647